CLINICAL TRIAL: NCT05644002
Title: A Puff Topography Biofeedback Paradigm to Reduce Stress-Precipitated Smoking Reinforcement
Brief Title: Puff Biofeedback to Reduce Smoking Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Teresa M. Leyro, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2020000645; R21DA052723 (NIH)
Record Dates: First submitted 2022-07-12; First posted 2022-12-09 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cigarette Smoking
Keywords: Smoking; Cigarette; Stress; Distress
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Sham Comparator): In this condition, participants are instructed to smoke as usual while attending to control stimuli presented to them on a computer monitor.
  Interventions: Behavioral: Control
- Puff Topography Biofeedback Training (PTBT) (Experimental): In this condition, participants are provided instructions on how to puff their cigarette via a computer-assisted paradigm.
  Interventions: Behavioral: Puff Topography Biofeedback Training

INTERVENTIONS:
Behavioral: Puff Topography Biofeedback Training — Visit 1: Participants will be asked to smoke their usual brand cigarette using the CReSS smoking topography device. Participants will be instructed on how to follow visual and auditory puffing prompts provided to them by a computer program in order to control puffing behavior for a duration of five minutes.
  Visit 2: Participants will be instructed to smoke their cigarette using the CReSS device and instructions provided during Visit 1 after undergoing a brief laboratory stress induction.
  Arms: Puff Topography Biofeedback Training (PTBT)
Behavioral: Control — Visit 1: Participants will be instructed to smoke their usual brand cigarette using the CReSS smoking topography device while passively viewing time-matched control stimulus presented to them on a computer monitor for a duration of five minutes.
  Visit 2: Participants will be instructed to smoke their cigarette using the CReSS device and instructions provided during Visit 1 after undergoing a brief laboratory stress induction.
  Other Names: Attention Control
  Arms: Control

SUMMARY:
The purpose of the study is to examine the effects of a novel bio-behavioral paradigm, entitled, Puff Topography Biofeedback Training, compared to a control condition, in reducing stress-induced smoking reinforcement.

DETAILED DESCRIPTION:
Smokers with emotional distress are particularly vulnerable to smoking reinforcement due to various biopsychological factors that contribute to deficits in emotion regulation and heightened reward processing, which undermine cessation efforts. Differences in puffing behavior may correspond with changes in cardiorespiratory parameters that may promote self-regulation and reduce craving.

This study is a between-subjects experimental test of Puff Topography Biofeedback Training (PTBT) and its ability to modify puff topography and cardiorespiratory activity during stress-precipitated smoking, and in turn, reduce acute smoking reinforcement.

Participants will be randomized to either PTBT or a Control condition and will complete two smoking trials on two successive days. The first smoking trial (Visit 1) will allow participants to gain familiarity with the task. The second smoking trial (Visit 2) will be completed following acute laboratory stress induction (stress-precipitated smoking trial).

The primary study aims are to test the effect of PTBT vs. Control as assessed via acute changes in stress-precipitated smoking reinforcement and changes in puffing behavior and cardiorespiratory parameters.The results of this high pre-intervention study could inform the subsequent development of a novel intervention strategy for improving quit outcomes in a treatment-resistant population.

The primary study aims are to test the effect of PTBT vs. Control in terms of: (a) objective puff topography parameters; (b) subjective reinforcement; and (c) whether physiological indices reflective of smoking reinforcement differ between conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Daily smoking ≥ 8 cigarettes/day verified by carbon monoxide analysis of breath sample ≥ 8 ppm
* Smoking within 30 minutes of waking
* English fluency.

Exclusion Criteria:

* Current smoking cessation treatment
* Past-month reduction of cigarettes/day by ≥50%
* Moderate or severe non-nicotine substance use disorder
* Past-year psychiatric instability (e.g., psychosis, mania)
* Severe visual, hearing, or cognitive impairments
* Medical condition that could impact stress reactivity or physiology
* Current regular use of medication that could affect cardiorespiratory function (e.g., beta blockers, benzodiazepines; note-use of SSRIs/SNRIs is permitted if dose is stable ≥ 6 wks).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Leyro, PhD, Principal Investigator — Rutgers, The State University of New Jersey; Samantha Farris, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers. The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data that underlie the primary study aims after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication of primary study aims. Ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically and theoretically sound proposal that is not redundant with the primary aims or findings already reported

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the greater Rutgers, New Brunswick community via posters in the local community and online advertisements. The first participant was enrolled on March 21, 2022, and the last participant was enrolled on September 8th 2023
Pre-assignment Details: The study involved one virtual session (Visit 0) at which preliminary eligibility was determined. 154 individuals consented at this virtual session. 90 participants were preliminarily eligible, and arrived at the subsequent first in person visit. 6 individuals were found to be ineligible at this session (e.g., biochemical verification of smoking status through expired carbon monoxide). In total 84 individuals were randomized to one of the two conditions in Visit 1.
Groups:
- Control: In this condition, participants are instructed to smoke as usual while attending to control stimuli presented to them on a computer monitor.
  Control: Visit 1: Participants will be instructed to smoke their usual brand cigarette using the CReSS smoking topography device while passively viewing time-matched control stimulus presented to them on a computer monitor for a duration of five minutes.
  Visit 2: Participants will be instructed to smoke their cigarette using the CReSS device and instructions provided during Visit 1 after undergoing a brief laboratory stress induction.
- Puff Topography Biofeedback Training (PTBT): In this condition, participants are provided instructions on how to puff their cigarette via a computer-assisted paradigm.
  Puff Topography Biofeedback Training: Visit 1: Participants will be asked to smoke their usual brand cigarette using the CReSS smoking topography device. Participants will be instructed on how to follow visual and auditory puffing prompts provided to them by a computer program in order to control puffing behavior for a duration of five minutes.
  Visit 2: Participants will be instructed to smoke their cigarette using the CReSS device and instructions provided during Visit 1 after undergoing a brief laboratory stress induction.
Period: Overall Study
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Started | 41 | 43
Finished Visit 1 | 41 | 43
Began Visit 2 | 40 | 40
Completed | 40 | 40
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who consented, were eligible, enrolled, were randomized, and completed both study visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.025 (7.427) | 40.950 (9.367) | 40.988 (8.399)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 22 | 26 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 12
  Not Hispanic or Latino | 38 | 30 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 28 | 28 | 56
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Purchase Task- Omax
Description: The Short-Cigarette Purchase Task (CPT) will be used to assess smoking reinforcement in response to stress-precipitated smoking. The CPT is based on progressive-ratio operant schedules wherein participants self-report their hypothetical cigarette consumption at various levels of price. Hypothetical purchasing will be based on the "last cigarette smoked". Five key behavioral economic indices of demand can be obtained from the CPT. One index reported here is the Omax, which is the number of cigarettes the individual endorses that they would purchase at the peak expenditure for a cigarette (i.e., highest endorsed US dollar per cigarette cost; Pmax).
Time Frame: Second Training Day following the Stress-Induction and Intervention (Smoking Task) i.e. post intervention, average 1 day.
Population: Participants who consented, were eligible, enrolled, were randomized, and completed both study visits. Four participants randomized randomized to the PTBT condition were removed due to being <80% adherent to the breathing/puff intervention prescribed, resulting in n=76 participants. An additional n=8 were excluded from these analyses due to invalid cigarette purchase task data resulting in a total of n=68 participants.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 36 | 32
cigarettes | 18.84 (23.96) | 18.80 (21.81)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction Omax between the PTBT and Control conditions; Test type: Other; p = .71, t-test, 2 sided — The threshold for statistical significance was p<.05; Levene's test for equal variances was used. If significance is <.05, equal variances are not assumed and reported results are adjusted accordingly; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [-9.09 to 13.21]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction Omax between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; degrees freedom = 66; t-statistic = 0.369
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 1, analysis 1]; Test type: Other; t-test, 2 sided; Hedge's g = .09

2. Primary Outcome: Modified Cigarette Evaluation Questionnaire - Cigarette Satisfaction Subscale
Description: The Modified Cigarette Evaluation Questionnaire (mCEQ) will be used to assess subjective smoking reinforcement. The mCEQ is a self-report measure that assesses how respondents feel about the "last cigarette smoked" with three subscales. One subscale indexes liking, or cigarette satisfaction. Score on this subscale range from 1 to 7, with higher scores reflecting greater subjective smoking satisfaction. Scores on the mCEQ cigarette satisfaction subscale administered post stress-precipitated smoking, during Visit 2, will be compared between conditions.
Time Frame: Second Training Day following the Stress-Induction and Intervention (Smoking Task) i.e. post intervention, average 1 days.
Population: Participants who consented, were eligible, enrolled, were randomized, and completed both study visits, Four participants randomized to the PTBT condition were removed due to being <80% adherent to the breathing/puff intervention prescribed, and an additional one participant was excluded from this analysis due to invalid mCEQ data, resulting in a total of n=75 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 39 | 36
score on a scale | 5.02 (1.68) | 5.27 (1.77)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction mCEQ cigarette satisfaction between the PTBT and Control conditions; Test type: Other; p = .530, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .251, 95% CI 2-sided [-.543 to 1.046]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 2, analysis 1]; Test type: Other; t-test, 2 sided; degrees freedom = 73; t-statistic = 0.631
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction mCEQ cigarette satisfaction between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; Hedge's g = .14

3. Primary Outcome: Cigarette Purchase Task - Intensity
Description: The Short-Cigarette Purchase Task (CPT) will be used to assess smoking reinforcement in response to stress-precipitated smoking. The CPT is based on progressive-ratio operant schedules wherein participants self-report their hypothetical cigarette consumption at various levels of price. Hypothetical purchasing will be based on the "last cigarette smoked". Five key behavioral economic indices of demand can be obtained from the CPT. One index reported here is intensity, which is the number of cigarettes consumed at zero cost.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 36 | 32
cigarettes | 13.86 (8.51) | 14.75 (8.11)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress intensity between the PTBT and Control conditions; Test type: Other; p = .66, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .889, 95% CI 2-sided [-3.149 to 4.927]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction intensity between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; degrees of freedom = 66; t-statistic = 0.439
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction intensity between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; Hedge's g = -.11

4. Primary Outcome: Cigarette Purchase Task- Pmax
Description: The Short-Cigarette Purchase Task (CPT) will be used to assess smoking reinforcement in response to stress-precipitated smoking. The CPT is based on progressive-ratio operant schedules wherein participants self-report their hypothetical cigarette consumption at various levels of price. Hypothetical purchasing will be based on the "last cigarette smoked". Five key behavioral economic indices of demand can be obtained from the CPT. One index reported here is the Pmax, which is the price at maximum expenditure for a cigarette.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: US dollars per cigarette
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 36 | 32
US dollars per cigarette | 5.07 (9.93) | 4.37 (8.61)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction Pmax between the PTBT and Control conditions; Test type: Other; p = .77, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.698, 95% CI 2-sided [-5.443 to 4.046]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction Pmax between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; degrees freedom = 66; t-statistic = -0.294
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 4, analysis 1]; Test type: Other; t-test, 2 sided; Hedge's g = -.071

5. Primary Outcome: Cigarette Purchase Task- Breakpoint
Description: The Short-Cigarette Purchase Task (CPT) will be used to assess smoking reinforcement in response to stress-precipitated smoking. The CPT is based on progressive-ratio operant schedules wherein participants self-report their hypothetical cigarette consumption at various levels of price. Hypothetical purchasing will be based on the "last cigarette smoked". Five key behavioral economic indices of demand can be obtained from the CPT. One index reported here is the breakpoint, which is the cost whereby consumption is suppressed to zero.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: US dollars per cigarette
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 36 | 32
US dollars per cigarette | 8.85 (11.82) | 8.50 (11.93)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction breakpoint between the PTBT and Control conditions; Test type: Other; p = .90, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.354, 95% CI 2-sided [-6.009 to 5.300]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction breakpoint between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; degrees of freedom = 66; t-statistic = -0.125
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 5, analysis 1]; Test type: Other; t-test, 2 sided; Hedge's g = -.03

6. Primary Outcome: Modified Cigarette Evaluation Questionnaire - Craving Reduction Subscale
Description: The Modified Cigarette Evaluation Questionnaire (mCEQ) will be used to assess subjective smoking reinforcement. The mCEQ is a self-report measure that assesses how respondents feel about the "last cigarette smoked" with three subscales. One subscale indexes wanting, or cigarette craving reduction. Score on this subscale range from 1 to 7, with higher scores reflecting greater subjective cigarette craving reduction. Scores on the mCEQ craving reduction subscale administered post stress-precipitated smoking, during Visit 2, will be compared between conditions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 39 | 36
units on a scale | 5.692 (1.575) | 4.944 (2.069)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction mCEQ craving reduction between the PTBT and Control conditions; Test type: Other; p = .09, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.748, 95% CI 2-sided [-1.601 to .105]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 6, analysis 1]; Test type: Other; t-test, 2 sided; degrees freedom = 65.261; t-statistic = -1.750
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction mCEQ craving reduction between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; Hedge's g = -.405

7. Primary Outcome: Modified Cigarette Evaluation Questionnaire - Psychological Reward Subscale
Description: The Modified Cigarette Evaluation Questionnaire (mCEQ) will be used to assess subjective smoking reinforcement. The mCEQ is a self-report measure that assesses how respondents feel about the "last cigarette smoked" with three subscales. One subscale indexes learning, or psychological reward. Score on this subscale range from 1 to 7, with higher scores reflecting greater subjective psychological reward. Scores on the mCEQ psychological reward subscale administered post stress-precipitated smoking, during Visit 2, will be compared between conditions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 39 | 36
units on a scale | 4.144 (1.768) | 4.328 (1.911)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress induction mCEQ psychological reward between the PTBT and Control conditions; Test type: Other; p = .666, t-test, 2 sided — The threshold for statistical significance was p<.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .184, 95% CI 2-sided [-.663 to 1.031]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 7, analysis 1]; Test type: Other; t-test, 2 sided; degrees freedom = 73; t-statistic = 0.184
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction mCEQ psychological reward between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; Hedge's g = .099

8. Secondary Outcome: Changes in Cardiac Vagal Control
Description: Beat-to-beat electrocardiograph and continuous respiration data were acquired using Thought Technology during the adaptation period and stress-precipitated smoking period. The data were and cleaned and scored using Mindware. Using Mindware, the IBI series is transformed to a heart period time series and then a heart power spectrum that is tapered using a Hamming window and finally a Fast Fourier Transform. Respiration data are similarly transformed using a Fast Fourier Transform to obtain a respiration power spectrum, and can be used to confirm the validity of the heart power spectrum data. Respiratory sinus arrhythmia is defined as variability in heart rate occurring in the high-frequency range, defined as 0.1 to 0.15 Hz corresponding with a respiratory rate between nine and 24 breaths per minute.
Time Frame: Second Training Day prior to Stress-Induction, and following Stress-Induction during Intervention (Smoking Task), average 1 day.
Population: Participants who consented, were eligible, enrolled, were randomized, and completed both study visits. Four participants randomized to the PTBT condition were removed due to being <80% adherent to the training, resulting in n=76 participants.
Measure: Mean (Standard Deviation); unit: milliseconds squared
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 40 | 36
milliseconds squared | 4.916 (1.380) | 4.778 (1.506)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); A multiple linear regression test was conducted to examine whether the PTBT intervention (versus control) significantly predicted post-stress-induction respiratory sinus arrhythmia during smoking, while controlling for average baseline respiratory sinus arrhythmia at step 1 of the model; Test type: Other; p = .73, Regression, Linear — The threshold for statistical significance was p<.05; Coding: Control=0, PTBT=1; β = .026, 95% CI 2-sided [-.358 to .507]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); A multiple linear regression test was conducted to examine whether the PTBT intervention (versus control) significantly predicted post-stress induction respiratory sinus arrhythmia during smoking, while controlling for average baseline respiratory sinus arrythmia at step 1 of the model; Test type: Other; Regression, Linear; degrees freedom = (2, 73); t-statistic = 0.345 — Condition (0=control; 1=PTBT)

9. Secondary Outcome: Puff Topography
Description: Puff topography indices will be objectively measured with the CReSS micro (Plowshare Technologies, Borgwaldt KC, Inc), a hand-held device that has a sterilized flow meter mouthpiece that is connected to a pressure transducer, which converts pressure into a digital signal that is sampled at 1,000Hz. Average Puff duration (sec) will be used to assess mechanism engagement from PTBT.
Time Frame: Second Training Day following Stress-Induction during Intervention (Smoking Task), average 1 day.
Population: Participants who consented, were eligible, enrolled, were randomized, and completed both study visits. Four participants randomized to the PTBT (active) condition were removed due to being <80% adherent to the breathing/puff intervention prescribed, resulting in n=76 participants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
Number analyzed (Participants) | 40 | 36
seconds | 2.05 (0.61) | 1.51 (0.38)
Statistical Analysis 1: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent samples t-test was conducted to examine differences in post-stress-induction average puff duration between PTBT and Control conditions; Test type: Other; p = .001, t-test, 2 sided — The threshold for statistical significance was p<.05; Levene's test for equal variances was used. If significance is < .05, equal variances are not assumed and reported results are adjusted accordingly; Mean Difference (Final Values) = -.543, 95% CI 2-sided [-.772 to -.314]
Statistical Analysis 2: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); [analysis description as in outcome 9, analysis 1]; Test type: Other; t-test, 2 sided; degrees freedom = 66.03; t-statistic = -4.739
Statistical Analysis 3: Comparison: Control vs Puff Topography Biofeedback Training (PTBT); An independent-samples t-test was conducted to examine differences in post-stress-induction average puff duration between the PTBT and Control conditions; Test type: Other; t-test, 2 sided; Hedge's g = -1.05

ADVERSE EVENTS:
Time Frame: Baseline (Visit 0; virtual preliminary eligibility assessment session), Visit 1, and Visit 2 (within four weeks from Visit 0).
Arm/Group | Control | Puff Topography Biofeedback Training (PTBT)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT05644002/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT05644002/ICF_001.pdf